CLINICAL TRIAL: NCT06679452
Title: Emotion, Aging and Forgiveness: Protocol of a Feasibility and Acceptability Study of Emotion-Focused Therapy for Older Individuals
Brief Title: Emotion, Aging, and Forgiveness: Protocol for a Feasibility of Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Bernardo Almeida, Dr, University Institute of Maia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University Maia
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Emotion-Focused Therapy; Aging; Forgiveness
Keywords: Emotion-Focused Therapy; Forgiveness; Aging; Randomized Controlled Trial; Feasibility Protocol
MeSH Terms: interventions — Emotion-Focused Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 35 participants randomly assigned to the EFT intervention (Experimental): The research will include 35 individuals aged 65 years or older, of both genders, who meet the study's inclusion criteria. Therapy sessions will be conducted individually and in person, in offices suited for psychological practice. Participants residing in senior housing will have the option, subject to agreement with their institution, to have sessions conducted in their facilities. Each session will last one hour and occur weekly over a three-month period, resulting in a total of 12 sessions per participant, in accordance with the EFT protocol for resolving emotional injuries established by Meneses and Greenberg (2019) and adjusted for this population/purposes by Almeida and Cunha (2024);
  Interventions: Other: Emotion-Focused Therapy
- 35 participants include in a control group (CG). (No Intervention): 35 participants included in a control group (CG), in the form of a waitlist.

INTERVENTIONS:
Other: Emotion-Focused Therapy — This feasibility protocol is a two-arm, parallel, double-blinded, RCT aimed at informing a future trial assessing the effectiveness of EFT in resolving emotional injuries in older adults in the context of interpersonal offenses.
  Arms: 35 participants randomly assigned to the EFT intervention

SUMMARY:
Over recent decades, Emotion-Focused Therapy, aging, and forgiveness have garnered significant attention in the field of psychology. However, there is a lack of studies on Emotion-Focused Therapy and forgiveness specifically tailored for older adults. This article describes a protocol to assess the feasibility and acceptability of a Randomized Controlled Trial of Emotion-Focused Therapy for the resolution of emotional injury in individuals over the age of 65 in the context of interpersonal offenses. The study is structured as a two-arm, parallel-group randomized trial with a waiting list control. We propose recruiting a sample of 70 participants, randomly assigned to either an immediate intervention group, which will receive Emotion-Focused Therapy over twelve weekly sessions, or a control group that will receive the same therapy after a twelve-week waiting period. Data will be collected in the beginning, middle, and at the end of therapy, and in two planned follow-ups (three and six months after therapy). Once this protocol is implemented, if the therapy proves to be feasible, acceptable, and shows promising results, the findings will inform a large-scale randomized clinical trial to advance the understanding of psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Our eligibility criteria include being 65 years or older, having experienced an interpersonal offense, residing at home or in a senior residence, stable prescribed medication use, scoring ≥ 26 on the MoCA (Montreal Cognitive Assessment), and fluency in Portuguese or English.

Exclusion Criteria:

* Exclusion criteria include reporting an offense which is less than a year old, severe emotional injuries (such as being a victim of domestic violence or abuse), psychiatric disorders, suicidal ideation, parasuicidal behavior, recent loss of a loved one, involvement in other therapies or clinical studies, current alcohol or drug abuse, living with another participant, and frequent hospitalizations.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Enright Forgiveness Inventory-EFI | From enrollment to the end of treatment at 12 weeks
  EFI is a self-report measure designed to measure the level of forgiveness in response to a specific offense. The EFI consists of 60 items divided into three 20-item subscales that assess affect, behavior, and cognition related to forgiveness, using a 6-point Likert scale. Scores range from 60 to 360, with higher scores indicating higher levels of forgiveness.
Letting Go (assessed through the Letting Go Measure; Greenberg et al., 2008): | From enrollment to the end of treatment at 12 weeks
  The Letting Go is a self-report instrument comprising a single item that evaluates the extent to which individuals have released their negative emotions toward the injurer. Responses are measured on a Likert scale ranging from 1 to 5.
The Unfinished Business Feelings and Needs Scale (UFB FN-Greenberg et al., 2008;) | From enrollment to the end of treatment at 12 weeks
  The Unfinished Business Feelings and Needs Scale (UFB FN-Greenberg et al., 2008; Singh, 1994) consists of a 6-item scale designed to measure the extent to which an individual who has experienced an unfair situation feels acceptance and empathy toward the person who has harmed them, utilizing a 5-point Likert scale.

SECONDARY OUTCOMES:
The European Portuguese World Health Organization Quality of Life Assessment in Older Adults (WHOQOL-OLD) | From enrollment to the end of treatment at 12 weeks
  The European Portuguese World Health Organization Quality of Life Assessment in Older Adults (WHOQOL-OLD) (Power et al., 2005; Vilar et al., 2016) comprises 28 items classified on a five-point scale and encompassing seven domains: sensory, autonomy, activities, social, death, intimacy, and family life (Vilar et al., 2016).
The Geriatric Depression Scale-15 (GDS-15; Matos et al., 2019; Yesavage & Sheikh, 1986) | From enrollment to the end of treatment at 12 weeks
  The Geriatric Depression Scale-15 (GDS-15; Matos et al., 2019; Yesavage & Sheikh, 1986) is specifically designed for screening depressive symptoms in older adults. It consists of 15 straightforward questions, each requiring a simple Yes or No response. The scale ranges from zero (indicating no depressive symptoms) to 15 points (representing the highest severity of depressive symptoms), with each affirmative response scored as 1 point. The cut-off points are defined as follows: 0 to 4 for the absence of depressive symptoms, 5 to 8 for mild symptoms, 9 to 11 for moderate symptoms, and 12 to 15 for severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Cunha Alexandra Dr, PhD, Study Chair — University of Maia
Locations (1):
- Av. Carlos Oliveira Campos - Castelo da Maia 4475-690 Avioso S. Pedro, Maia, Castelo Da Maia, Portugal

REFERENCES:
- [Background] Buzgova R, Kozakova R, Bobcikova K, Zelenikova R. Predictors of life satisfaction in elders living at home in the Czech Republic. PLoS One. 2023 Mar 30;18(3):e0283772. doi: 10.1371/journal.pone.0283772. eCollection 2023. PMID 36996129
- [Background] Lopez J, Serrano MI, Gimenez I, Noriega C. Forgiveness Interventions for Older Adults: A Review. J Clin Med. 2021 Apr 26;10(9):1866. doi: 10.3390/jcm10091866. PMID 33925790
- [Background] Band-Winterstein T, Eisikovits Z, Brownell P, King A. Introduction: exploring older women's perspectives on lifetime abuse. J Elder Abuse Negl. 2024; 36(2):91-92. 10.1080/08946566.2024.2332141.
- [Background] Toussaint LL, Worthington EL, Williams DR, eds. Forgiveness and Health: Scientific Evidence and Theories Relating Forgiveness to Better Health. Springer; 2015. doi: 10.1007/978-94-017-9993-5.
- [Background] Greenberg LJ, Warwar SH, Malcolm WM. Differential effects of Emotion-Focused Therapy and psychoeducation in facilitating forgiveness and letting go of emotional injuries. J Couns Psychol. 2008; 55(2):185-96. doi: 10.1037/0022-0167.55.2.185.
- [Background] Almeida, B., Cunha, C. Time, resentment, and forgiveness: Impact on the well-being of older adults. Trends in Psychology. 2023. https://doi.org/10.1007/s43076-023-00343-2
- [Background] Enright RD, Fitzgibbons RP. Forgiveness therapy: An empirical guide for resolving anger and restoring hope. American Psychological Association; 2015. doi: 10.1037/14526-000.
- [Background] Meneses CW, Greenberg LS. Forgiveness and letting go in Emotion-Focused Therapy. American Psychological Association; 2019. doi: 10.1037/0000144-000.
- [Background] Worthington EL, Wade NG, eds. Handbook of forgiveness. 2nd ed. Routledge; 2020.
- See also: The present study explores how resentment and forgiveness can affect older people and how resentment can be alleviated or intensified over time. The investigation is based on a qualitative methodology, using life history interviews, carried out in two mo — https://doi.org/10.1007/s43076-023-00343-2